CLINICAL TRIAL: NCT02459990
Title: Congenital Malformations and Maternal Use of Anti-hypertensive Medication in the United Kingdom
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2452R00003
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: Hypertension malformation fetal mortality
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assess Fetal Mortality and Malformations in Women treated with antihypertensive medication during preganancy. Mother - Child pairs will be analysed in a cohort selected from the UK in the CPRD database. Years covered are 1997 to 2014. Aim is to assess the risk of Antihypertensive treatment in women.

DETAILED DESCRIPTION:
Women with chronic hypertension are at risk of experiencing severe complications such as adverse effects of fetal growth, survival, and renal function during pregnancy. General recommendations advocate the treatment of high blood pressure during pregnancy to decrease these risks to the mother and child, with extreme caution. Many studies assessing the risk of congenital malformations in infants whose mothers were treated with anti-hypertensive medication have been inconclusive, in part due to the variability of the original data sources and possibly the robustness of the analyses.2 Studies regarding this health issue have been unable to stratify anti-hypertensive medications sufficiently to truly assess the risk per drug class, Angiotensin II Receptor Antagonists/Blockers (ARBs) and Angiotensin-converting-enzyme inhibitor (ACE inhibitor) in particular.We will attempt to assess the prescription rate of ARBs and ACE inhibitors among women with very high blood pressure in the United Kingdom (UK) and estimate the risk of serious foetal outcomes in women treated with ARBs and/or ACEs and who may also have the following co-morbid conditions: Diabetes Types I or II, Diabetic Nephropathy, and Congestive Heart Failure.

ELIGIBILITY:
Inclusion Criteria: age and gender -

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who may become pregnant ages 18-50 in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incident cases of Fetal Mortality among hypertensive women | up to 17 years
  Number of incident Fetal mortality cases among hypertensive women, study period duration is 204 months (start date 1997 to end of follow-up date 2014)
Incident cases of Fetal Malformation among hypertensive women | up to 17 years
  Number of incident Fetal Malformation cases among hypertensive women, study period duration is 204 months (start date 1997 to end of follow-up date 2014)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3810&filename=Synopsis.pdf